CLINICAL TRIAL: NCT03535467
Title: Caregiver Burden in Stroke: Robot-Assisted Therapy vs Conventional Rehabilitation
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif GÜLER, Principal Investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREH1
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Stroke Rehabilitation and Caregivers
Keywords: Caregivers; Exoskeleton Device; Stroke Rehabilitation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Rehabilitation
  Interventions: Other: Caregiver's Burden Inventory
- Robotic Therapy
  Interventions: Other: Caregiver's Burden Inventory

INTERVENTIONS:
Other: Caregiver's Burden Inventory — The Caregiver Burden Inventory was developed by Canadian researchers.The authors of the instrument stress the importance of using a multidimensional measurement of burden with separate scores for each dimension in as opposed to global or uni-dimensional scores.

SUMMARY:
Caregiver's burden in rehabilitation is important for both patients physical and mental health. Therefore researching caregivers burden and treatment of any depression or associated any psychological disorders of caregiver is crucial.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia after stoke, Brunnstrom stages: stage 2-3 of lower limb minimum 6 months after stroke,

Exclusion Criteria:

* More than 1 stroke, aphasia, Dysphagia, other life life threatening diseases Independent ambulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-65 years old stroke patients who are not ambulatuar and dependent to their caregivers.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden Inventory | 15 days
  Caregiver Burden Inventory(CBI) first designed by Novak and Guest in 1989 to measure burden of patient's caregiver. Caregiver can be a relative or a professional. CBI consists of 5 different subscales(Time Dependency Items(5 question),Development Items(5 question),Physical Health Items(4 question),Emotional Health Items(5 question),Social Relationship Items(5 question)), a total of 24 questions. Every question should be answered by the caregiver according to a likert scale (0=Never,1=Rarely,2=Sometimes,3=Quite Frequently,4=Nearly Always) and a total of 96 points. 36 point is a limit to a professional help for caregiver and the higher the points get there is more burden for caregiver.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Taksim Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guler MA, Erhan B, Yilmaz Yalcinkaya E. Caregiver burden in stroke inpatients: a randomized study comparing robot-assisted gait training and conventional therapy. Acta Neurol Belg. 2021 Jun;121(3):729-736. doi: 10.1007/s13760-020-01465-5. Epub 2020 Aug 10. PMID 32776169